CLINICAL TRIAL: NCT06036732
Title: The New Developed FIVE Score and Its Comparison With GCS and FOUR Scores Regarding Length of Hospital Stay Morbidity and Mortality in Neuro-intensive Care Patients. an Observational Prospective Study
Brief Title: A New Approach in Intensive Care Unit Consciousness Assessment: FIVE Score
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, merve tugba ozfidan donmez, medical doctor, Istanbul University - Cerrahpasa
Other Study IDs: E-72109855-604.01.01-7591
Record Dates: First submitted 2023-04-27; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Postoperative Intracranial Hematoma; Postoperative Intracranial Haemorrhage; Supratentorial Cancer; Infratentorial Neoplasms; Arnold Chiari Malformation; Subarachnoid Hemorrhage; Traumatic Brain Injury; Epilepsy, Temporal Lobe; Cerebrovascular Event; Intensive Care Neurological Disorder; Coma; Unconsciousness; Assessment, Self
Keywords: FIVE Score; FOUR Score; GCS; Modified Rankin Score; Neuro-ICU
MeSH Terms: conditions — Supratentorial Neoplasms; Infratentorial Neoplasms; Arnold-Chiari Malformation; Subarachnoid Hemorrhage; Brain Injuries, Traumatic; Epilepsy, Temporal Lobe; Coma; Unconsciousness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. The primary aim of this study is to investigate the correlation between the length of ICU stay and a newly developed FIVE score in neuro-intensive care patients.
2. The secondary objectives are to evaluate the impact of the FIVE score on hospital length of stay, Modified Rankin Scale, and mortality, as well as to determine the correlation between the GCS, FOUR, and FIVE scores

DETAILED DESCRIPTION:
Consciousness monitoring is crucial in neuro-intensive care. Despite the use of different scoring systems to establish a common language among evaluators, the Glasgow Coma Scale (GCS) remains the most widely used in clinical practice. In GCS evaluation, verbal response, motor response, and eye response are assessed. Another scoring system, FOUR (Full Outline of UnResponsiveness ) Score is similar to the Glasgow Coma Score (GCS). But it is designed to provide a more comprehensive neurological assessment. The FOUR score evaluates four areas: including eye opening, motor response, brainstem reflexes, and respiration, and assigns a score for each area. A comprehensive education regarding those scores was given the intensive care healthcare providers before the trial.

In this study, the investigators developed the Full Intracranial Validity Evaluation (FIVE) Score, by adding the mean arterial pressure and gag reflex components to the FOUR score. The investigators believe that this new score, which can be used for clinical monitoring, may offer an alternative to FOUR and GCS monitoring. According to this scoring system, in addition to the criteria for the FOUR score, patients with a mean arterial pressure between 60-130mmHg receive 2 points; patients under inotropic support with a mean arterial pressure between 60-130mmHg receive 1 point; patients with a mean arterial pressure below 60mmHg or above 130mmHg receive 0 points. Additionally, for patients with infratentorial mass, the investigators add the assessment of gag reflex in the calculation of the FIVE score. If the reflex is absent, 0 points are given; if it is unilateral, 1 point is given, and if it is preserved, 2 points are given.

The demographic data, diagnoses, systemic comorbidities, the American Society of Anaesthesiologists (ASA) score, the Charlson Comorbidity Index (CCI), and the APACHE II scores of patients were recorded.

The GCS, FOUR, and FIVE scores of the patients were recorded at neuro ICU admission, every 12 hours during neuro ICU follow-up period and discharge. In our clinic, GCS monitoring is routinely performed hourly for every patient admitted to the ICU. For patients with a decrease of two or more points in GCS score, FOUR and FIVE scores were re-evaluated and recorded without waiting for the 12 hours. Besides this, the worst, the best and the mean GCS, FOUR, and FIVE scores were recorded in the neuro ICU follow-up period. The assessment count of the GCS, FOUR, and FIVE scores during clinical follow-up was recorded.

The length of ICU and hospital stay were recorded. The Modified Rankin Scale of the patients was recorded six months after ICU discharge.

The primary aim of this study is to investigate the correlation between the length of ICU stay and a newly developed FIVE score in neuro-intensive care patients. The secondary objectives are to evaluate the impact of the FIVE score on length of hospital stay, Modified Rankin Scale, and mortality, as well as to determine the correlation between the GCS, FOUR, and FIVE scores.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18 and 80
* who were monitored in the Neurosurgical Intensive Care Unit
* had a history of ischemic or hemorrhagic stroke within the last 6 months
* underwent infratentorial craniotomy
* supratentorial craniotomy
* endoscopic surgery
* vascular surgery
* epilepsy surgery
* hydrocephalus surgery
* neurovascular intervention

Exclusion Criteria:

* patients over 80 years of age
* under 18 years of age
* patients who were sedated
* patients who were administered neuromuscular blockers during intensive care follow-up
* patients with diagnosed psychiatric illness
* patients who were alcohol or drug addicts

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients between the ages of 18 and 80, who were monitored in the Neurosurgical Intensive Care Unit and had a history of ischemic or hemorrhagic stroke within the last 6 months, underwent infratentorial craniotomy, supratentorial craniotomy, endoscopic surgery, vascular surgery, epilepsy surgery, hydrocephalus surgery, or neurovascular intervention, were included in the study
Sampling Method: Non-Probability Sample
Enrollment: 223 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-01-25 (Estimated); Study Completion 2024-02-25 (Estimated)

PRIMARY OUTCOMES:
Change in FIVE Scores | baseline, 12 hours intervals, up to an hour of ICU discharge
  Full Intracranial Validity Evaluation, minimum value:0, maximum value: 20, higher scores mean a better situation
Change in GKS Scores | baseline, 12 hours intervals, up to an hour of ICU discharge
  Glasgow Coma Score, minimum value:3, maximum value: 15, higher scores mean a better situation
Modified Rankin Scale | six months after ICU discharge
  In scoring post-discharge morbidity six months after intensive care unit discharge, Modified Rankin Score is used. minimum value:0, maximum value:6, higher scores mean a worse outcome

OTHER OUTCOMES:
Length of stay in ICU | From hospitalization to hospital discharge, estimated average = 10 days
  Length of neuro ICU follow-up period
Length of stay in hospital | From hospitalization to hospital discharge, estimated average = 10 days
  Length of hospital follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Korkmaz Dilmen, MD, Study Chair — Istanbul University - Cerrahpasa; Yusuf Tunali, MD, Study Director — Istanbul University - Cerrahpasa; Fatma Eren Akcil, MD, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University- Cerrahpasa(IUC), Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Glasgow Coma Scale (GCS) and Four/Five Scores, along with the highest, lowest, and average scores, discharge scores, Modified Rankin Scores at 6 months post-discharge, and length of stay information measured upon admission to the intensive care unit will be shared.